CLINICAL TRIAL: NCT01277211
Title: A Randomized, Open-Label, Controlled, Multi-Center Trial to Evaluate the Contraceptive Efficacy, Cycle Control, Safety and Acceptability of NuvaRing® (SCH 900702) in Chinese Women
Brief Title: A Study to Evaluate the Effectiveness of NuvaRing® to Prevent Pregnancies in Chinese Women (P06450)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P06450
Record Dates: First submitted 2011-01-12; First posted 2011-01-14 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2024-06-20 (Actual); Status verified 2022-02

CONDITIONS: Contraception
Keywords: Contraception; NuvaRing
MeSH Terms: interventions — Endoglin; NuvaRing; drospirenone; drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ENG-EE (NuvaRing) (Experimental): Participants were to complete 13 cycles of etonogestrel (ENG) and ethinylestradiol (EE) use. Each cycle was 28 days, with a 21-day active treatment period followed by a 7-day ring-free period. Participants used one ring per cycle. Each ring contained 11.7 mg ENG and 2.7 mg EE, and released on average 120 mcg/day of ENG and 15 mcg/day of EE.
  Interventions: Drug: ENG 120 µg + EE 15 µg intravaginal ring
- DRSP-EE (Active Comparator): Participants were to complete 13 cycles of drospirenone (DRSP) and ethinylestradiol (EE) use. Each cycle was 28 days, with a 21-day active treatment period followed by a 7-day tablet-free period. Participants received a total of 21 tablets of DRSP-EE per cycle. Each tablet contained 3 mg DRSP and 30 μg EE.
  Interventions: Drug: DRSP 3 mg + EE 30 µg

INTERVENTIONS:
Drug: ENG 120 µg + EE 15 µg intravaginal ring — 13 cycles of ENG-EE (NuvaRing) vaginal ring use. Each cycle 28 days, with a 21-day active treatment period followed by 7-day ring-free period. One ring per cycle, each ring containing 11.7 mg ENG and 2.7 mg EE, and releasing on average 120 mcg/day of ENG and 15 mcg/day of EE.
  Other Names: NuvaRing
  Arms: ENG-EE (NuvaRing)
Drug: DRSP 3 mg + EE 30 µg — 13 cycles of DRSP-EE tablet use. Each cycle 28 days, with a 21-day active treatment period followed by a 7-day tablet-free period. Participants received total of 21 tablets per cycle, each tablet contained 3 mg DRSP and 30 μg EE.
  Other Names: Yasmin
  Arms: DRSP-EE

SUMMARY:
This is a study to assess the effectiveness of NuvaRing® (SCH 900702) for the prevention of pregnancy in fertile Chinese women. The acceptability and safety of NuvaRing® will also be assessed and compared with that of Yasmin.

DETAILED DESCRIPTION:
The purpose of this study is to assess the contraceptive efficacy of NuvaRing in fertile Chinese women; to assess vaginal bleeding pattern (cycle control), general safety, and acceptability of NuvaRing; and to evaluate the NuvaRing's effect on dysmenorrhea.

ELIGIBILITY:
Key Inclusion Criteria:

* Sexually active Chinese women, at risk for pregnancy and not planning to use condoms during trial medication use
* Women in need for contraception and willing to use a hormonal contraceptive method for 13 cycles
* Body mass index ≥18 and ≤29 kg/m^2

Key Exclusion Criteria:

* Contraindications for contraceptive steroids
* Abnormal cervical smear corresponding to indeterminate changes at screening
* Clinically relevant abnormal laboratory result at screening as judged by the investigator.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 983 (Actual)
Dates: Start 2011-09-19 (Actual); Primary Completion 2013-09-18 (Actual); Study Completion 2013-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fan GS, Ren M, Di W, Su P, Chang Q, Wu S, Qin Y, Korver T, Marintcheva-Petrova M, Yacik C, McCrary Sisk C, Wang G. Efficacy and safety of the contraceptive vaginal ring (NuvaRing) compared with a combined oral contraceptive in Chinese women: a 1-year randomised trial. Eur J Contracept Reprod Health Care. 2016 Aug;21(4):303-9. doi: 10.1080/13625187.2016.1186269. Epub 2016 Jun 24. PMID 27339759

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 983 participants randomized, 946 received treatment and 37 discontinued prior to receiving treatment.
Period: Overall Study
Arm/Group | ENG-EE (NuvaRing) | DRSP-EE
Started | 738 | 245
Treated | 714 | 232
Completed | 588 | 182
Not Completed | 150 | 63
Not completed — Adverse Event | 60 | 22
Not completed — Pregnancy | 9 | 4
Not completed — Lost to Follow-up | 14 | 9
Not completed — Did not wish to continue | 17 | 0
Not completed — Withdrew Consent | 9 | 9
Not completed — Non-compliance with protocol | 13 | 4
Not completed — Did not meet protocol eligibility | 1 | 0
Not completed — Administrative | 3 | 0
Not completed — Pregnancy wish | 0 | 2
Not completed — Discontinued prior to treatment | 24 | 13

BASELINE CHARACTERISTICS:
Population: All Subjects Treated (AST) group, which consisted of all randomized participants who used at least one ring/pill.
Groups:
- Total: Total of all reporting groups
Arm/Group | ENG-EE (NuvaRing) | DRSP-EE | Total
Number analyzed (Participants) | 714 | 232 | 946
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.8 (4.0) | 31.2 (3.9) | 31.7 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 714 | 232 | 946
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pearl Index, by Treatment Group
Description: Primary Efficacy Outcome measure for this study was contraceptive efficacy, or the prevention of in-treatment pregnancy. The total incidence of in-treatment pregnancies was expressed as the Pearl Index, which is defined as the number of in-treatment pregnancies per 100 woman-years of exposure (one woman-year defined as a period of 365.25 days).
Time Frame: Up to 1 year
Population: Restricted Intent-to-Treat (R-ITT) Group, which consisted of all participants from the Intent-to-Treat (ITT) Group who had at least one cycle at risk (no condom use and confirmed intercourse).
Measure: Mean (95% Confidence Interval); unit: Pregnancies per 100 woman-years
Arm/Group | ENG-EE (NuvaRing) | DRSP-EE
Number analyzed (Participants) | 662 | 216
Pregnancies per 100 woman-years | 1.92 [0.92 to 3.53] | 3.12 [1.01 to 7.29]
Statistical Analysis 1: Comparison: ENG-EE (NuvaRing) vs DRSP-EE; Differences between the two treatment groups (ENG-EE vs. DRSP-EE) were explored using an exact 95% CI for the Ratio of the two Pearl Indices based on the Poisson distribution; Test type: Superiority or Other; p = 0.531, Poisson distribution method; Differences between treatment groups was explored using an exact 95% CI for the ratio of the two Pearl Indices based on the Poisson distribution; Ratio of Pearl Indices = 0.61, 95% CI 2-sided [0.19 to 2.29]

2. Secondary Outcome: Percentage of Participants With Intermenstrual (Breakthrough) Bleeding/Spotting, by Cycle
Description: Participants kept diaries to record vaginal bleeding events. They were asked to record, on a daily basis, whether they experienced vaginal bleeding, which included BLEEDING or SPOTTING, at any time during a cycle other than normal menstruation while in the study. (This is also known as "breakthough" bleeding.) Vaginal bleeding that required >=2 pads/tampons per day was classified as BLEEDING. Vaginal bleeding that required <=1 pad/tampon per day was classified as SPOTTING.
Time Frame: Up to 1 year
Population: ITT Group, which consisted of all randomized participants who used at least one ring/pill.
Measure: Number; unit: Percentage of participants
Arm/Group | ENG-EE (NuvaRing) | DRSP-EE
Number analyzed (Participants) | 714 | 232
Percentage of participants
  Cycle 1 (n=598,199) | 18.6 [15.5 to 21.9] | 21.6 [16.1 to 28.0]
  Cycle 2 (n=604,195) | 12.3 [9.7 to 15.1] | 18.5 [13.3 to 24.6]
  Cycle 3 (n=578,196) | 8.5 [6.3 to 11.1] | 14.3 [9.7 to 20.0]
  Cycle 4 (n=587,194) | 7.5 [5.5 to 9.9] | 15.5 [10.7 to 21.3]
  Cycle 5 (n=592,187) | 6.8 [4.9 to 9.1] | 8.0 [4.6 to 12.9]
  Cycle 6 (n=590,185) | 6.9 [5.0 to 9.3] | 10.8 [6.7 to 16.2]
  Cycle 7 (n=583,186) | 7.5 [5.5 to 10.0] | 11.3 [7.1 to 16.7]
  Cycle 8 (n=585,188) | 6.3 [4.5 to 8.6] | 10.6 [6.6 to 16.0]
  Cycle 9 (n=576,187) | 6.9 [5.0 to 9.3] | 8.0 [4.6 to 12.9]
  Cycle 10 (n=572,183) | 5.9 [4.2 to 8.2] | 10.4 [6.4 to 15.7]
  Cycle 11 (n=578,177) | 4.2 [2.7 to 6.1] | 7.9 [4.4 to 12.9]
  Cycle 12 (n=569,176) | 5.3 [3.6 to 7.4] | 9.7 [5.7 to 15.0]
  Cycle 13 (n=544,173) | 6.4 [4.5 to 8.8] | 11.0 [6.7 to 16.6]
Statistical Analysis 1: Comparison: ENG-EE (NuvaRing) vs DRSP-EE; For Cycle 1, a two-sided 95% CI for the difference in percentage between the treatment groups (ENG-EE vs. DRSP-EE) was calculated using the method of Miettinen and Nurminen; Test type: Superiority or Other; p = 0.346, Miettinen and Nurminen method; Difference in Percentages, Cycle 1 = -3.0, 95% CI 2-sided [-9.9 to 3.1]
Statistical Analysis 2: Comparison: ENG-EE (NuvaRing) vs DRSP-EE; For Cycle 2, a two-sided 95% CI for the difference in percentage between the treatment groups (ENG-EE vs. DRSP-EE) was calculated using the method of Miettinen and Nurminen; Test type: Superiority or Other; p = 0.029, Miettinen and Nurminen method; Difference in Percentages, Cycle 2 = -6.2, 95% CI 2-sided [-12.7 to -0.6]
Statistical Analysis 3: Comparison: ENG-EE (NuvaRing) vs DRSP-EE; For Cycle 3, a two-sided 95% CI for the difference in percentage between the treatment groups (ENG-EE vs. DRSP-EE) was calculated using the method of Miettinen and Nurminen; Test type: Superiority or Other; p = 0.019, Miettinen and Nurminen method; Difference in Percentages, Cycle 3 = -5.8, 95% CI 2-sided [-11.8 to -0.9]
Statistical Analysis 4: Comparison: ENG-EE (NuvaRing) vs DRSP-EE; For Cycle 4, a two-sided 95% CI for the difference in percentage between the treatment groups (ENG-EE vs. DRSP-EE) was calculated using the method of Miettinen and Nurminen; Test type: Superiority or Other; p = 0.001, Miettinen and Nurminen method; Difference in Percentages, Cycle 4 = -8.0, 95% CI 2-sided [-14.0 to -2.9]
Statistical Analysis 5: Comparison: ENG-EE (NuvaRing) vs DRSP-EE; For Cycle 5, a two-sided 95% CI for the difference in percentage between the treatment groups (ENG-EE vs. DRSP-EE) was calculated using the method of Miettinen and Nurminen; Test type: Superiority or Other; p = 0.556, Miettinen and Nurminen method; Difference in Percentages, Cycle 5 = -1.3, 95% CI 2-sided [-6.4 to 2.6]
Statistical Analysis 6: Comparison: ENG-EE (NuvaRing) vs DRSP-EE; For Cycle 6, a two-sided 95% CI for the difference in percentage between the treatment groups (ENG-EE vs. DRSP-EE) was calculated using the method of Miettinen and Nurminen; Test type: Superiority or Other; p = 0.089, Miettinen and Nurminen method; Difference in Percentages, Cycle 6 = -3.9, 95% CI 2-sided [-9.5 to 0.5]
Statistical Analysis 7: Comparison: ENG-EE (NuvaRing) vs DRSP-EE; For Cycle 7, a two-sided 95% CI for the difference in percentage between the treatment groups (ENG-EE vs. DRSP-EE) was calculated using the method of Miettinen and Nurminen; Test type: Superiority or Other; p = 0.110, Miettinen and Nurminen method; Difference in Percentages, Cycle 7 = -3.7, 95% CI 2-sided [-9.4 to 0.8]
Statistical Analysis 8: Comparison: ENG-EE (NuvaRing) vs DRSP-EE; For Cycle 8, a two-sided 95% CI for the difference in percentage between the treatment groups (ENG-EE vs. DRSP-EE) was calculated using the method of Miettinen and Nurminen; Test type: Superiority or Other; p = 0.049, Miettinen and Nurminen method; Difference in Percentages, Cycle 8 = -4.3, 95% CI 2-sided [-9.8 to -0.0]
Statistical Analysis 9: Comparison: ENG-EE (NuvaRing) vs DRSP-EE; For Cycle 9, a two-sided 95% CI for the difference in percentage between the treatment groups (ENG-EE vs. DRSP-EE) was calculated using the method of Miettinen and Nurminen; Test type: Superiority or Other; p = 0.621, Miettinen and Nurminen method; Difference in Percentages, Cycle 9 = -1.1, 95% CI 2-sided [-6.2 to 2.9]
Statistical Analysis 10: Comparison: ENG-EE (NuvaRing) vs DRSP-EE; For Cycle 10, a two-sided 95% CI for the difference in percentage between the treatment groups (ENG-EE vs. DRSP-EE) was calculated using the method of Miettinen and Nurminen; Test type: Superiority or Other; p = 0.041, Miettinen and Nurminen method; Difference in Percentages, Cycle 10 = -4.4, 95% CI 2-sided [-10.0 to -0.2]
Statistical Analysis 11: Comparison: ENG-EE (NuvaRing) vs DRSP-EE; For Cycle 11, a two-sided 95% CI for the difference in percentage between the treatment groups (ENG-EE vs. DRSP-EE) was calculated using the method of Miettinen and Nurminen; Test type: Superiority or Other; p = 0.046, Miettinen and Nurminen method; Difference in Percentages, Cycle 11 = -3.8, 95% CI 2-sided [-8.9 to -0.1]
Statistical Analysis 12: Comparison: ENG-EE (NuvaRing) vs DRSP-EE; For Cycle 12, a two-sided 95% CI for the difference in percentage between the treatment groups (ENG-EE vs. DRSP-EE) was calculated using the method of Miettinen and Nurminen; Test type: Superiority or Other; p = 0.037, Miettinen and Nurminen method; Difference in Percentages, Cycle 12 = -4.4, 95% CI 2-sided [-9.9 to -0.2]
Statistical Analysis 13: Comparison: ENG-EE (NuvaRing) vs DRSP-EE; For Cycle 13, a two-sided 95% CI for the difference in percentage between the treatment groups (ENG-EE vs. DRSP-EE) was calculated using the method of Miettinen and Nurminen; Test type: Superiority or Other; p = 0.048, Miettinen and Nurminen method; Difference in Percentages, Cycle 13 = -4.5, 95% CI 2-sided [-10.4 to -0.0]

3. Secondary Outcome: Percentage of Participants With Absence of Withdrawal Bleeding, by Cycle
Description: Participants kept diaries to record vaginal bleeding events. They were asked to record, on a daily basis, whether vaginal bleeding was present. Absence of withdrawal bleeding was defined as no bleeding/spotting during the expected bleeding period.
Time Frame: Up to 1 year
Population: ITT Group, which consisted of all randomized participants who used at least one ring/pill.
Measure: Number; unit: Percentage of participants
Arm/Group | ENG-EE (NuvaRing) | DRSP-EE
Number analyzed (Participants) | 714 | 232
Percentage of participants
  Cycle 1 (n=596,199) | 8.6 [6.4 to 11.1] | 14.6 [10.0 to 20.3]
  Cycle 2 (n=602,195) | 4.8 [3.2 to 6.8] | 9.7 [6.0 to 14.8]
  Cycle 3 (n=577,196) | 5.2 [3.5 to 7.3] | 11.7 [7.6 to 17.1]
  Cycle 4 (n=586,194) | 4.1 [2.6 to 6.0] | 7.7 [4.4 to 12.4]
  Cycle 5 (n=590,187) | 5.4 [3.7 to 7.6] | 6.4 [3.4 to 10.9]
  Cycle 6 (n=588,185) | 5.8 [4.0 to 8.0] | 9.7 [5.9 to 14.9]
  Cycle 7 (n=581,186) | 3.4 [2.1 to 5.3] | 7.5 [4.2 to 12.3]
  Cycle 8 (n=583,188) | 5.0 [3.4 to 7.1] | 6.9 [3.7 to 11.5]
  Cycle 9 (n=575,187) | 4.3 [2.8 to 6.4] | 8.6 [5.0 to 13.5]
  Cycle 10 (n=571,183) | 3.7 [2.3 to 5.6] | 6.6 [3.4 to 11.2]
  Cycle 11 (n=576,177) | 3.0 [1.7 to 4.7] | 7.3 [4.0 to 12.2]
  Cycle 12 (n=568,176) | 4.0 [2.6 to 6.0] | 10.2 [6.2 to 15.7]
  Cycle 13 (n=543,173) | 5.9 [4.1 to 8.2] | 10.4 [6.3 to 15.9]
Statistical Analysis 1: Comparison: ENG-EE (NuvaRing) vs DRSP-EE; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.015, Miettinen and Nurminen method; Difference in Percentages, Cycle 1 = -6.0, 95% CI 2-sided [-12.0 to -1.1]
Statistical Analysis 2: Comparison: ENG-EE (NuvaRing) vs DRSP-EE; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.012, Miettinen and Nurminen method; Difference in Percentages, Cycle 2 = -4.9, 95% CI 2-sided [-10.1 to -1.0]
Statistical Analysis 3: Comparison: ENG-EE (NuvaRing) vs DRSP-EE; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.002, Miettinen and Nurminen method; Difference in Percentages, Cycle 3 = -6.5, 95% CI 2-sided [-12.0 to -2.2]
Statistical Analysis 4: Comparison: ENG-EE (NuvaRing) vs DRSP-EE; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.044, Miettinen and Nurminen method; Difference in Percentages, Cycle 4 = -3.6, 95% CI 2-sided [-8.5 to -0.1]
Statistical Analysis 5: Comparison: ENG-EE (NuvaRing) vs DRSP-EE; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.609, Miettinen and Nurminen method; Difference in Percentages, Cycle 5 = -1.0, 95% CI 2-sided [-5.7 to 2.5]
Statistical Analysis 6: Comparison: ENG-EE (NuvaRing) vs DRSP-EE; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.062, Miettinen and Nurminen method; Difference in Percentages, Cycle 6 = -3.9, 95% CI 2-sided [-9.3 to 0.2]
Statistical Analysis 7: Comparison: ENG-EE (NuvaRing) vs DRSP-EE; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; p = 0.019, Miettinen and Nurminen method; Difference in Percentages, Cycle 7 = -4.1, 95% CI 2-sided [-9.0 to -0.6]
Statistical Analysis 8: Comparison: ENG-EE (NuvaRing) vs DRSP-EE; [analysis description as in outcome 2, analysis 8]; Test type: Superiority or Other; p = 0.308, Miettinen and Nurminen method; Difference in Percentages, Cycle 8 = -1.9, 95% CI 2-sided [-6.7 to 1.6]
Statistical Analysis 9: Comparison: ENG-EE (NuvaRing) vs DRSP-EE; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.027, Miettinen and Nurminen method; Difference in Percentages, Cycle 9 = -4.2, 95% CI 2-sided [-9.3 to -0.4]
Statistical Analysis 10: Comparison: ENG-EE (NuvaRing) vs DRSP-EE; [analysis description as in outcome 2, analysis 10]; Test type: Superiority or Other; p = 0.098, Miettinen and Nurminen method; Difference in Percentages, Cycle 10 = -2.9, 95% CI 2-sided [-7.6 to 0.5]
Statistical Analysis 11: Comparison: ENG-EE (NuvaRing) vs DRSP-EE; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p = 0.009, Miettinen and Nurminen method; Difference in Percentages, Cycle 11 = -4.4, 95% CI 2-sided [-9.4 to -1.0]
Statistical Analysis 12: Comparison: ENG-EE (NuvaRing) vs DRSP-EE; [analysis description as in outcome 2, analysis 12]; Test type: Superiority or Other; p = 0.002, Miettinen and Nurminen method; Difference in Percentages, Cycle 12 = -6.2, 95% CI 2-sided [-11.7 to -2.1]
Statistical Analysis 13: Comparison: ENG-EE (NuvaRing) vs DRSP-EE; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.043, Miettinen and Nurminen method; Difference in Percentages, Cycle 13 = -4.5, 95% CI 2-sided [-10.2 to -0.1]

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | ENG-EE (NuvaRing) | DRSP-EE
Serious Adverse Events (participants affected / at risk) | 2/714 | 4/232
Other Adverse Events (participants affected / at risk) | 0/714 | 0/232
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ENG-EE (NuvaRing) (N=714) | DRSP-EE (N=232)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review and comment on data analysis and presentation for all abstracts, manuscripts, and slide presentations that report any results of this trial 45 days prior to the submission for publication or presentation.